CLINICAL TRIAL: NCT04391751
Title: Basal Joint Arthroplasty and Carpal Tunnel Release Comparing Single Versus Double Incision. Randomized Clinical Trial
Brief Title: Concomitant Basal Joint Arthroplasty and Carpal Tunnel Release
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(ATR)147/2018
Record Dates: First submitted 2020-04-29; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Carpal Tunnel Syndrome; Osteoarthritis Thumb
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single incision (Experimental): Carpal tunnel release and basal joint arthroplasty through a single radial approach
  Interventions: Procedure: Carpal tunnel release and basal joint arthroplasty through single incision
- Double incision (Active Comparator): Double approach: carpal tunnel release through palmar approach and basal joint arthroplasty through radial approach
  Interventions: Procedure: Carpal tunnel release and basal joint arthroplasty through double incision

INTERVENTIONS:
Procedure: Carpal tunnel release and basal joint arthroplasty through single incision — Group I: experimental - single incision The surgical technique chosen for thumb basal join was trapeziectomy with ligamentous reconstruction and tendon interposition (LRTI), using flexor carpi radialis (FCR). Through a dorsal approach over trapeziometacarpal joint, the entire trapezium was excised. Volar traction of FCR allowed us to longitudinally incise the deep leaflet of FCR tendon until flexor pollicis longus (FPL) tendon was clearly visualized. Then, ulnar half of FCR tendon was harvested proximally through a second transverse incision in middle third of the forearm and split all the way to its insertion on the index metacarpal. A hole was placed in the base of the first metacarpal and FCR tendon was routed through the bone canal and then fixed with non-reabsorbable sutures. Finally, the tendon remanent was rolled up and placed into the trapezial void to act as a spacer.
  Arms: Single incision
Procedure: Carpal tunnel release and basal joint arthroplasty through double incision — Group II: active comparator - double incision Trapezial excision and ligament reconstruction were performed in the same way as in group I, except that FCR deep leaflet was not incised. After radial incision wound closure, carpal tunnel release was performed through a second separate longitudinal palmar incision.
  Arms: Double incision

SUMMARY:
Concomitant carpal tunnel syndrome and basal thumb junt osteoarthritis through a single incision has been described. Case serials have reported good with this technique. Nonetheless, there is a lack of comparative studies evaluating the effectivity and complications of single-incision versus double-incision technique. Only with an randomized clinical trial design it is possible to gain evidence about the advantages of one treatment method over another. The aim of the study is the comparison between two surgical techniques for concomitant carpal tunnel syndrome and basal thumb junt osteoarthritis: single versus double incision techniques.

DETAILED DESCRIPTION:
Basal thumb joint osteoarthritis is a common disorder especially among postmenopausal women. In this specific subgroup of patients, radiographic signs appear in up to 40%.

Approximately 28% of those cases are symptomatic. Its pathoanatomy and treatment has been well described. Trapeziometacarpal joint is the most commonly joint requiring treatment for osteoarthritis in the upper extremity, often involving removing the trapezius. The same demographic group is also frequently affected by carpal tunnel syndrome (CTS), which coexists with basal joint arthritis in 18% to 46% of patients. In those cases, a combined surgical approach has been reported to be beneficial. The two conditions have traditionally been treated surgically through separate incisions.

a radial incision for trapeziectomy and standard midline volar carpal tunnel incision for median nerve decompression. Trapeziectomy has been proved to provide some degree of carpal tunnel decompression. However, as previous studies have suggested, release of the transverse carpal ligament should be performed in addition to basal joint arthroplasty incision, as trapeziectomy by itself does not completely decompress the carpal tunnel. The ability to decompress the carpal tunnel during basal joint arthroplasty using a single incision would allow to shorten surgery time, improve appearance, and potentially decrease morbidity compared to a staged or two-incision procedure. We sought to determine whether carpal tunnel release using a single incision during basal joint arthroplasty is as effective as two-incision approach in patients with concomitant CTS and basal thumb joint osteoarthrosis. The secondary hypothesis is that single incision prevents from morbidity associated to a second incision, such as pillar pain, longer surgical procedure, infection rate or necrosis of the skin bridge between incisions

ELIGIBILITY:
Inclusion Criteria:

* Concomitant basal joint osteoarthritis and CTS in the ipsilateral extremity.
* Severe CTS sympthoms wiht positive physical examination findings (eg, Phalen test and Tinel test).
* Electromyography (EMG) results supporting the diagnosis of CTS.
* Failed CTS nonsurgical treatment.
* Basal joint osteoarthritis Eaton stage II or greater
* Unacceptable pain localized in the basal joint appeared with activity, or reproduced by grind test or direct palpation
* Failed basal joint osteoarthritis nonsurgical treatment.

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus
* Acute trauma
* Rheumatoid arthritis
* Hipothyroidism
* Hyperthiroidism
* Posttraumatic arthritis
* Prior hand surgery procedures
* Nerve compression at proximal level
* Other nerve entrapments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of CTS symptoms intensity | Preoperatively, 3, 6, and 12 months postoperatively
  To assess the CTS symptoms intensity, patients filled out the Boston Carpal Tunnel Questionaire. This questionnaire evaluates symptom's severity (11 items) and functional status (8 items) (1: no complaints, 5 maximum complaints possible).
  Minimum score is 19 and maximum 95.

SECONDARY OUTCOMES:
Change of hand function | Preoperatively, 3, 6, and 12 months postoperatively
  Hand function was assessed through Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH). Minimum score is 0 (no disability) and maximum 100 (total disability).
Change of hand pain | Preoperatively, 3, 6, and 12 months postoperatively
  Pain was assessed through 10-visual analog scale. Minimum score is 0 (no pain) and maximum 10 (sever pain).
Change of grip strength | Preoperatively, 3, 6, and 12 months postoperatively
  Grip strength was measured the mean of 3 attempts, in kilograms, with correction for hand dominance, using a standard dynamometer.

OTHER OUTCOMES:
Complications associated with the different surgical procedures | At 2 weeks posteoperatively
  Complications such as pillar pain, longer surgical procedure, infection rate or necrosis of the skin bridge between incisions

CONTACTS AND LOCATIONS:
Locations (1):
- Ignacio Esteban Feliu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton RI, Pellegrini VD Jr. Surgical management of basal joint arthritis of the thumb. Part II. Ligament reconstruction with tendon interposition arthroplasty. J Hand Surg Am. 1986 May;11(3):324-32. doi: 10.1016/s0363-5023(86)80137-x. PMID 3711604
- [Background] Eaton RG, Lane LB, Littler JW, Keyser JJ. Ligament reconstruction for the painful thumb carpometacarpal joint: a long-term assessment. J Hand Surg Am. 1984 Sep;9(5):692-99. doi: 10.1016/s0363-5023(84)80015-5. PMID 6491213
- [Background] Weiss AC, Goodman AD. Thumb Basal Joint Arthritis. J Am Acad Orthop Surg. 2018 Aug 15;26(16):562-571. doi: 10.5435/JAAOS-D-17-00374. PMID 29969109
- [Background] Armstrong AL, Hunter JB, Davis TR. The prevalence of degenerative arthritis of the base of the thumb in post-menopausal women. J Hand Surg Br. 1994 Jun;19(3):340-1. doi: 10.1016/0266-7681(94)90085-x. PMID 8077824
- [Background] Geoghegan JM, Clark DI, Bainbridge LC, Smith C, Hubbard R. Risk factors in carpal tunnel syndrome. J Hand Surg Br. 2004 Aug;29(4):315-20. doi: 10.1016/j.jhsb.2004.02.009. PMID 15234492
- [Background] Lutsky K, Ilyas A, Kim N, Beredjiklian P. Basal joint arthroplasty decreases carpal tunnel pressure. Hand (N Y). 2015 Sep;10(3):403-6. doi: 10.1007/s11552-014-9724-9. PMID 26330770
- [Background] Cassidy C, Glennon PE, Stein AB, Ruby LK. Basal joint arthroplasty and carpal tunnel release through a single incision: an in vitro study. J Hand Surg Am. 2004 Nov;29(6):1085-8. doi: 10.1016/j.jhsa.2004.07.003. PMID 15576220
- [Background] Ingari JV, Romeo N. Basal Joint Arthroplasty and Radial-sided Carpal Tunnel Release Using a Single Incision. Tech Hand Up Extrem Surg. 2015 Dec;19(4):157-60. doi: 10.1097/BTH.0000000000000100. PMID 26422193
- [Derived] Esteban-Feliu I, Gallardo-Calero I, Barrera-Ochoa S, Vidal-Tarrason N, Mir X, Lluch-Bergada A. Basal joint arthroplasty and carpal tunnel release comparing a single versus double incision: a prospective randomized study. Eur J Orthop Surg Traumatol. 2022 Oct;32(7):1391-1397. doi: 10.1007/s00590-021-03086-x. Epub 2021 Sep 22. PMID 34550476